CLINICAL TRIAL: NCT06998498
Title: Prehabilitation for Aortic Aneurysm Surgery: Proof-of-concept Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Celano, Associate Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025P001463
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Aortic Aneurysm
Keywords: Aortic aneurysm; Prehabilitation; Collaborative care
MeSH Terms: conditions — Aortic Aneurysm | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ready for Recovery (Experimental): Participants in this arm will receive the Ready for Recovery intervention.
  Interventions: Behavioral: Ready for Recovery

INTERVENTIONS:
Behavioral: Ready for Recovery — The Ready for Recovery program is a 6-week, multicomponent, tailored, prehabilitation intervention to promote the optimization of medical and psychological status prior to surgery. Its key components include education, enhancement of beneficial health behaviors, reduction of negative psychological symptoms, and the promotion of social support. Following an initial session, the team will develop a customized prehabilitation plan for each participant. Participants will work towards goals each week and will discuss progress with their study trainer via weekly phone sessions, which will continue until the scheduled surgical procedure.

SUMMARY:
This is a single-arm, proof-of-concept trial to examine the feasibility, acceptability, and preliminary efficacy of the Ready for Recovery program, a 6-week collaborative care intervention to help prepare individuals for repair of aortic aneurysms.

DETAILED DESCRIPTION:
This is a single-arm, proof-of-concept trial to examine the feasibility, acceptability, and preliminary efficacy of the Ready for Recovery program. Ready for Recovery is a 6-week collaborative care program to prepare individuals for surgical procedures to repair an aortic aneurysm. Participants will speak with a study trainer on the phone each week and will set goals related to physical activity, a healthy diet, and inspiratory muscle training. They also will be given resources to reduce stress, treat anxiety and depression (if present), and stop smoking, and the study team will make recommendations regarding medication adjustments to reduce complications after surgery. The primary outcome is feasibility (measured by percentage of phone sessions completed). Secondary outcomes include acceptability (measured by weekly 0-10 utility ratings) and preliminary impact on functional, psychological, and health behavior outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing elective aortic aneurysm repair (open or endovascular)

Exclusion Criteria:

* Cognitive disturbance
* Current pregnancy or plan to become pregnant prior to surgery
* Inability to write/speak fluently in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | Weekly over 6 weeks
  Percentage of intervention phone sessions completed

SECONDARY OUTCOMES:
Feasibility of data collection | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Proportion of assessment sessions in which outcome data is obtained from participants and the medical record
Utility of the Ready for Recovery program | 6 weeks
  Participants will rate the utility of the Ready for Recovery program on an 11-point Likert scale (0-10), with 0 being not at all helpful and 10 being very helpful.
Change in physical function (PROMIS PF-20) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Physical function will be measured using the 20-item PROMIS Physical Function Scale (PROMIS PF-20). PROMIS PF-20 scores range from 20 to 100, with higher scores indicating higher levels of physical function.

OTHER OUTCOMES:
Change in physical health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] physical component score) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  The SF-12 physical component score will be used to assess physical health-related quality of life (Range: 0-100). Higher scores indicate higher levels of physical health-related quality of life.
Change in mental health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] mental component score) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  The SF-12 mental component score will be used to assess mental health-related quality of life (Range: 0-100). Higher scores indicate higher levels of mental health-related quality of life.
Change in depressive symptoms (9-item Patient Health Questionnaire [PHQ-9]) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Depressive symptoms will be measured using the 9-item Patient Health Questionnaire (PHQ-9). The PHQ-9 ranges from 0-27, with higher scores indicating higher levels of depression.
Change in anxiety symptoms (7-item Generalized Anxiety Disorder Scale [GAD-7]) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Anxiety will be measured using the 7-item Generalized Anxiety Disorder scale (GAD-7). The GAD-7 ranges from 0-21, with higher scores indicating higher levels of anxiety
Change in perceived stress (Perceived Stress Scale) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Perceived stress will be assessed via the Perceived Stress Scale (PSS). PSS scores range from 0-40, with higher scores indicating higher levels of perceived stress.
Change in cognition (telephonic Montreal Cognitive Assessment [t-MoCA]) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Cognition will be measured using the telphonic Montreal Cognitive Assessment (t-MoCA). t-MoCA scores range from 0 to 22, with higher scores indicating better cognition.
Change in perceived social support (Multidimensional Scale of Perceived Social Support) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Perceived social support will be measured by the Multidimensional Scale of Perceived Social Support (MSPSS). MSPSS scores range from 1-7, with higher scores indicating higher levels of perceived social support.
Change in self-reported physical activity (International Physical Activity Questionnaire [IPAQ]; in metabolic equivalent-minutes/week) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  This will be measured via the International Physical Activity Questionnaire (IPAQ) as a secondary measure of physical activity.
Changes in cigarette smoking (in number of cigarettes smoked per week) | Baseline, post-intervention (1-5 days prior to surgery), post-operation (1-2 days before or after hospital discharge), 90 days post-discharge
  Participants will be asked how many cigarettes they have smoked in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No